CLINICAL TRIAL: NCT06869941
Title: Adipose Tissue Gene Expression and Metabolomics Links to the Gut Microbiome-brain Axis (POINSETTIA Study)
Brief Title: Adipose Tissue Gene Expression and Metabolomics Links to the Gut Microbiome-brain Axis
Acronym: POINSETTIA
Status: Recruiting | Type: Observational
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, José Manuel Fernández-Real, Principal investigator, clinical professor, section chief of Endocrinology and Nutrition Department of Josep Trueta University Hospital, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Other Study IDs: POINSETTIA-2024.200
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Continous Glucose Monitoring; Cognition; Gut-microbiota-brain axis
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — saliva, stool, blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OBESITY: With 2 subgroups
  * Man with obesity
  * Women with obesity
- WITHOUT OBESITY: With 2 subgroups:
  * Man without obesity
  * Women without obesity

SUMMARY:
This study aims to understand how adipose tissue (fat) and the gut microbiota (the bacteria in the gut) may influence brain function and cognition. It has been observed that changes in adipose tissue in animals such as mice and Drosophila (a type of insect) affect memory and other brain functions. Additionally, it is believed that the gut microbiota also plays an important role in cognition.

This study will explore how gene expression in adipose tissue, blood metabolites, and the gut microbiota are related to cognitive function, such as memory and thinking, in individuals with and without obesity. The investigation will also assess whether these factors can predict changes in the brain over time and how they influence sleep, physical activity, and blood sugar regulation.

Advanced technologies will be used to analyze samples of tissue, blood, and microbiota, with the goal of identifying new mechanisms through which obesity affects the brain. This research may contribute to the development of new diagnostic and therapeutic strategies for cognitive problems in individuals with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >20 years old.
* Scheduled for surgical intervention to extract adipose tissue.
* Signed informed consent for study participation.

Exclusion Criteria:

* Not meeting inclusion criteria.
* Non-obesity-related systemic diseases (cancer, severe kidney/liver disease).
* Systemic diseases with intrinsic inflammation (rheumatoid arthritis, Crohn's disease, asthma, chronic infections (HIV/tuberculosis)) or any type of infectious disease.
* Pregnant/breastfeeding women.
* Persons under legal/administrative restrictions.
* Those with infection symptoms in the past month.
* Use of antibiotics/antifungals/antivirals (previous 3 months).
* Chronic steroidal/anti-inflammatory drug use.
* Major psychiatric history.
* Excessive alcohol intake, acute or chronic (>40g/day (women), >80g/day (men)) or drug abuse.
* Immunosuppressants treatment.
* Participants with severe eating disorders.
* Serum liver enzymes (GOT, GPT) above twice the upper limit of normal. Obvious signs or symptoms of liver disease, acute or chronic hepatitis.
* History of iron balance disorders (e.g., genetic hemochromatosis, hemosiderosis from any cause, atransferrinemia, paroxysmal nocturnal hemoglobinuria).
* Creatinine greater than 1.2 and glomerular filtration rate below 40.
* Current treatment for malignant neoplasia, other than basal cell or squamous cell skin cancer.
* Heart disease classified as class III or IV, known ischemic cardiovascular disease.
* Renal failure, history of kidney transplant, or current dialysis treatment.
* Chronic constipation (bowel movement frequency ≥ 7 days) .

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will make use of the existing samples from the FATBANK cohort (a platform driven by CIBEROBN, managed by the IDIBGI Biobank, and part of the Spanish National Biobank Network). Participants in this cohort had previously signed informed consent to be contacted again. Therefore, the selected participants will be reappointed at the Endocrinology, Diabetes, and Nutrition Service (UDENTG) of the Dr. Josep Trueta Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Glycemic variability | 36 month
  Mean and standard deviation of glucose measures in mg/dL using a CGM 10 days.
The percentage of time in glucose target range (glucose level 100mg/dl-125mg/dl) | 36 months
The glycaemic risk measured with the low blood glucose index (LBGI) | 36 months
  Low blood glucose index (LBGI) is a parameter that quantifies the risk of glycaemic.
The glycaemic variability measured with mean amplitude of glycaemic excursions (MAGE) | 36 months
  measured in mg/dl
Minutes light sleep | 36 months
  Mean and standard deviation of minutes' light sleep measures by activity and sleep tracker device.
Minutes deep sleep | 36 months
  Mean and standard deviation of minutes' deep sleep measures by activity and sleep tracker device.
Minutes rapid eye movement (REM) | 36 months
  Mean and standard deviation of minutes REM measures by activity and sleep tracker device.

SECONDARY OUTCOMES:
Audioverbal memory | 36 months
  It will be measured by California Verbal Learning Test (CVLT). Minimum/maximum scale values (0-16), where 16 is a better audioverbal memory.
Effect on gut microbiota | 36 months
  Gut microbiota will be analysed by metagenomics and metabolomics.
Visual memory | 36 months
  It will be measured by Rey-Osterrieth Complex Figure. Minimum/maximum scale values (0-36), where 36 is a better visual memory.
Depressive symptomatology | 36 months
  It will be measured by Patient Health Questionnaire-9 (PHQ-9). Minimum/maximum scale values (0-27), where ≥ 20 is severe depression.
Impulsivity | 36 months
  It will be measured by Impulsive Behaviour Scale (UPPS-P). The test evaluates: Negative urgency (tendency to act rashly under extreme negative emotions), Lack of Premeditation (tendency to act without thinking), Lack of Perseverance (inability to remain focused on a task) and Sensation Seeking (tendency to seek out novel and thrilling experiences). All items are rated on a four point scale from 1 (strongly agree) to 4 (strongly disagree).
Food Addiction | 36 months
  It will be measured by Yale Food Addiction Scale. It is a symptom score from 0-11, based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria, for substance dependence. Food addiction is diagnosed if ≥3 symptoms are reported.
Behavioural inhibition | 36 months
  It will be measured by Sensitivity to Punishment and Sensitivity to Reward (SPSRQ). The scale of Sensitivity to Punishment is related to the behavioural inhibition system. It is made up of two subscales of 24 items each. For each subscale, the minimum score is 0 and the maximum score is 24, with higher scores indicating greater sensitivity to punishment or reward, respectively.
Behavioural activation | 36 months
  It will be measured by Sensitivity to Punishment and Sensitivity to Reward (SPSRQ). The reward sensitivity scale is related to the behavioural activation system. The questionnaire consists of two subscales of 24 items each. Each subscale ranges from 0 (minimum) to 24 (maximum), where a higher score indicates greater sensitivity to reward or punishment, respectively.
Visoconstructive function | 36 months
  It will be measured by Rey-Osterrieth Complex Figure. Minimum/maximum scale values (0-36), where 36 is a better visoconstructive function.
Selective and alternating attention | 36 months
  It will be measured by Trail making test (Part A and B).
Attention and working memory | 36 months
  It will be measured by the Digits subtest of the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV). This subtest includes two parts: Digits Forward (measuring attention) and Digits Backward (measuring working memory). The total raw score ranges from 0 (minimum) to 30 (maximum), with higher scores indicating better attention and working memory capacity.
Inhibition | 36 months
  It will be measured by Stroop Color-Word Test.
Phonemic verbal fluency | 36 months
  It will be measured by PMR.
Semantic verbal fluency | 36 months
  It will be measured by Animals test. The person must name as many animals as possible in 1 minute. The result is corrected by standard scores, according to age and level of education.
Facial recognition | 36 months
  It will be measured by Picture of Facial Recognition Test (POFA).
Emotion recognition | 36 months
  It will be measured by Benton Facial Recognition Test (BFRT). This test evaluates the recognition of the five basic emotions: happiness, sadness, surprise, disgust, and anger.
Binge eating disorder | 36 months
  It will be measured by Binge Eating Scale (BES). The BES is one of the most widely used measures to assess binge eating disorder symptomatology. The BES score ranges from 0 to 46 and its cut-off point is greater than or equal to 27. Subjects with scores higher than 27 are more likely to suffer from binge eating disorder.
Anxiety state | 36 months
  It will be measured by State-Trate Anxiety Inventory (STAI). This questionnaire evaluates state anxiety (S) and trait anxiety (R) through 20 items each, with a likert-type response scale of four alternatives. In the case of state anxiety, the scale goes from 0 (not at all) to 3 (a lot), while for trait anxiety it goes from 0 (almost never) to 3 (almost always). The higher the score, the greater the anxiety in both concepts.
Effect on brain structure | 36 months
  Brain structure will be assessed using magnetic resonance imaging.
Diffusion Tensor Imaging brain sequences | 36 months
  Diffusion Tensor Imaging was acquired at 1.5 T (Philips ingenia) using a single-shot spin echo sequence with echo-planar imaging (EPI), 50 contiguous slices, voxel size 2x2x2.5 mm3, TE/TR of 72/3581 ms/ms, a diffusion-weighting factor b = 800 s/mm2 and diffusion encoding along 32 directions.
Brain iron accumulation | 36 months
  It will be assessed using magnetic resonance imaging using (R2*)
Resting-state functional brain sequences | 36 months
  It will be assessed using magnetic resonance imaging (T2*-weighted echo-planar imaging). T2 * relaxation data will be acquired with a multi-echo gradient sequence with 10 equidistant echoes (first echo = 4.6ms; echo spacing = 4.6ms; repetition time = 1300ms). The value of T2 * will be calculated by adjusting the simple exponential terms for the signal decay of the respective echo time values.
Insulin resistance | 36 months
  It will be measured by HOMA
Markers of chronic inflammation (C-reactive protein, IL-6, adiponectin and soluble, tumour necrosis factor-α receptor fractions) | 36 months
  Enzyme-linked immunosorbent assay (ELISA) and quantitative polymerase chain reaction (qPCR)
Glycosylated haemoglobin (HbA1c) value | 36 months
  Glycosylated haemoglobin (HbA1c) in % or mmol/mol
The percentage of time in hyperglycaemia (glucose level above 250 mg/dl) | 36 months
The percentage of time in hypoglycaemia (glucose level below 70mg/dl) | 36 months
The percentage of time in glucose range (glucose level below 100 mg/dl) | 36 months
The percentage of time in glucose range (glucose level between 126-139 mg/dl) | 36 months
The percentage of time in glucose range (glucose level between 140-199 mg/dl) | 36 months
The percentage of time in glucose range (glucose level above 200 mg/dl) | 36 months
Burned calories | 36 months
  Mean and standard deviation of burned calories measures by activity and sleep tracker device.
Steps Mean and standard deviation of steps measures by activity and sleep tracker device. | 36 months
  The mean and standard deviation of steps refer to the average number of steps taken by a participant and how much those steps vary from the average, as measured by an activity and sleep tracker device. The mean is the average, while the standard deviation shows the variation or consistency in step count.
Distance Mean and standard deviation of distance measures by activity and sleep tracker device. | 36 months
Minutes null activity | 36 months
  Mean and standard deviation of minutes' null activity measures by activity and sleep
Minutes slight activity | 36 months
  Mean and standard deviation of minutes slight activity measures by activity and sleep
Minutes mean activity | 36 months
  Mean and standard deviation of minutes mean activity measures by activity and sleep tracker device.
Minutes high activity | 36 months
  Mean and standard deviation of minutes high activity measures by activity and sleep tracker device.
Calories | 36 months
  Mean and standard deviation of calories measures by activity and sleep tracker device.
Minutes asleep | 36 months
  Mean and standard deviation of minutes asleep measures by activity and sleep tracker.
Minutes awake | 36 months
  Mean and standard deviation of minutes awake measures by activity and sleep tracker.
Bed time Mean and standard deviation of bed time measures by activity and sleep tracker device. | 36 months
Number time awake Mean and standard deviation of number time awake measures by activity and sleep | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Fernández-Real, M.D., Ph.D., Principal Investigator — Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Locations (1):
- Institut d'Investigació Biomèdica de Girona (IDIBGI), Girona, Girona, Spain

REFERENCES:
- [Background] Mayneris-Perxachs J, Arnoriaga-Rodriguez M, Garre-Olmo J, Puig J, Ramos R, Trelis M, Burokas A, Coll C, Zapata-Tona C, Pedraza S, Perez-Brocal V, Ramio L, Ricart W, Moya A, Jove M, Sol J, Portero-Otin M, Pamplona R, Maldonado R, Fernandez-Real JM. Presence of Blastocystis in gut microbiota is associated with cognitive traits and decreased executive function. ISME J. 2022 Sep;16(9):2181-2197. doi: 10.1038/s41396-022-01262-3. Epub 2022 Jun 21. PMID 35729225
- [Background] Bier E. Drosophila, the golden bug, emerges as a tool for human genetics. Nat Rev Genet. 2005 Jan;6(1):9-23. doi: 10.1038/nrg1503. PMID 15630418
- [Background] Douglas AE. The Drosophila model for microbiome research. Lab Anim (NY). 2018 Jun;47(6):157-164. doi: 10.1038/s41684-018-0065-0. Epub 2018 May 23. PMID 29795158
- [Background] Quesada-Vazquez S, Castells-Nobau A, Latorre J, Oliveras-Canellas N, Puig-Parnau I, Tejera N, Tobajas Y, Baudin J, Hildebrand F, Beraza N, Burcelin R, Martinez-Gili L, Chilloux J, Dumas ME, Federici M, Hoyles L, Caimari A, Del Bas JM, Escote X, Fernandez-Real JM, Mayneris-Perxachs J. Potential therapeutic implications of histidine catabolism by the gut microbiota in NAFLD patients with morbid obesity. Cell Rep Med. 2023 Dec 19;4(12):101341. doi: 10.1016/j.xcrm.2023.101341. PMID 38118419
- [Background] Mayneris-Perxachs J, Moreno-Navarrete JM, Ballanti M, Monteleone G, Alessandro Paoluzi O, Mingrone G, Lefebvre P, Staels B, Federici M, Puig J, Garre J, Ramos R, Fernandez-Real JM. Lipidomics and metabolomics signatures of SARS-CoV-2 mediators/receptors in peripheral leukocytes, jejunum and colon. Comput Struct Biotechnol J. 2021;19:6080-6089. doi: 10.1016/j.csbj.2021.11.007. Epub 2021 Nov 8. PMID 34777716
- [Background] Lin H, Peddada SD. Analysis of compositions of microbiomes with bias correction. Nat Commun. 2020 Jul 14;11(1):3514. doi: 10.1038/s41467-020-17041-7. PMID 32665548
- [Background] Albanese D, Donati C. Strain profiling and epidemiology of bacterial species from metagenomic sequencing. Nat Commun. 2017 Dec 22;8(1):2260. doi: 10.1038/s41467-017-02209-5. PMID 29273717
- [Background] Zhao S, Li H, Han W, Chan W, Li L. Metabolomic Coverage of Chemical-Group-Submetabolome Analysis: Group Classification and Four-Channel Chemical Isotope Labeling LC-MS. Anal Chem. 2019 Sep 17;91(18):12108-12115. doi: 10.1021/acs.analchem.9b03431. Epub 2019 Sep 5. PMID 31441644
- [Background] Arnoriaga-Rodriguez M, Mayneris-Perxachs J, Burokas A, Contreras-Rodriguez O, Blasco G, Coll C, Biarnes C, Miranda-Olivos R, Latorre J, Moreno-Navarrete JM, Castells-Nobau A, Sabater M, Palomo-Buitrago ME, Puig J, Pedraza S, Gich J, Perez-Brocal V, Ricart W, Moya A, Fernandez-Real X, Ramio-Torrenta L, Pamplona R, Sol J, Jove M, Portero-Otin M, Maldonado R, Fernandez-Real JM. Obesity Impairs Short-Term and Working Memory through Gut Microbial Metabolism of Aromatic Amino Acids. Cell Metab. 2020 Oct 6;32(4):548-560.e7. doi: 10.1016/j.cmet.2020.09.002. PMID 33027674
- [Background] Mayneris-Perxachs J, Castells-Nobau A, Arnoriaga-Rodriguez M, Garre-Olmo J, Puig J, Ramos R, Martinez-Hernandez F, Burokas A, Coll C, Moreno-Navarrete JM, Zapata-Tona C, Pedraza S, Perez-Brocal V, Ramio-Torrenta L, Ricart W, Moya A, Martinez-Garcia M, Maldonado R, Fernandez-Real JM. Caudovirales bacteriophages are associated with improved executive function and memory in flies, mice, and humans. Cell Host Microbe. 2022 Mar 9;30(3):340-356.e8. doi: 10.1016/j.chom.2022.01.013. Epub 2022 Feb 16. PMID 35176247
- [Background] Mayneris-Perxachs J, Castells-Nobau A, Arnoriaga-Rodriguez M, Martin M, de la Vega-Correa L, Zapata C, Burokas A, Blasco G, Coll C, Escrichs A, Biarnes C, Moreno-Navarrete JM, Puig J, Garre-Olmo J, Ramos R, Pedraza S, Brugada R, Vilanova JC, Serena J, Gich J, Ramio-Torrenta L, Perez-Brocal V, Moya A, Pamplona R, Sol J, Jove M, Ricart W, Portero-Otin M, Deco G, Maldonado R, Fernandez-Real JM. Microbiota alterations in proline metabolism impact depression. Cell Metab. 2022 May 3;34(5):681-701.e10. doi: 10.1016/j.cmet.2022.04.001. PMID 35508109
- [Background] Oliveras-Canellas N, Castells-Nobau A, de la Vega-Correa L, Latorre-Luque J, Motger-Alberti A, Arnoriaga-Rodriguez M, Garre-Olmo J, Zapata-Tona C, Coll-Martinez C, Ramio-Torrenta L, Moreno-Navarrete JM, Puig J, Villarroya F, Ramos R, Casado-Anguera V, Martin-Garcia E, Maldonado R, Mayneris-Perxachs J, Fernandez-Real JM. Adipose tissue coregulates cognitive function. Sci Adv. 2023 Aug 11;9(32):eadg4017. doi: 10.1126/sciadv.adg4017. Epub 2023 Aug 11. PMID 37566655
- [Background] Xia D, Kelleher RJ 3rd, Shen J. Loss of Abeta43 Production Caused by Presenilin-1 Mutations in the Knockin Mouse Brain. Neuron. 2016 Apr 20;90(2):417-22. doi: 10.1016/j.neuron.2016.03.009. PMID 27100200
- [Background] Wechsler, D. WAIS IV: Escala de Inteligencia de Wechsler para Adultos-IV. Madrid: TEA. 2012
- [Background] Guo DH, Yamamoto M, Hernandez CM, Khodadadi H, Baban B, Stranahan AM. Beige adipocytes mediate the neuroprotective and anti-inflammatory effects of subcutaneous fat in obese mice. Nat Commun. 2021 Jul 30;12(1):4623. doi: 10.1038/s41467-021-24540-8. PMID 34330904
- [Background] Guo DH, Yamamoto M, Hernandez CM, Khodadadi H, Baban B, Stranahan AM. Visceral adipose NLRP3 impairs cognition in obesity via IL-1R1 on CX3CR1+ cells. J Clin Invest. 2020 Apr 1;130(4):1961-1976. doi: 10.1172/JCI126078. PMID 31935195
- [Background] Sodhi K, Pratt R, Wang X, Lakhani HV, Pillai SS, Zehra M, Wang J, Grover L, Henderson B, Denvir J, Liu J, Pierre S, Nelson T, Shapiro JI. Role of adipocyte Na,K-ATPase oxidant amplification loop in cognitive decline and neurodegeneration. iScience. 2021 Oct 12;24(11):103262. doi: 10.1016/j.isci.2021.103262. eCollection 2021 Nov 19. PMID 34755095
- [Background] Morrison SF, Nakamura K. Central Mechanisms for Thermoregulation. Annu Rev Physiol. 2019 Feb 10;81:285-308. doi: 10.1146/annurev-physiol-020518-114546. Epub 2018 Sep 26. PMID 30256726
- [Background] Cardoso F, Klein Wolterink RGJ, Godinho-Silva C, Domingues RG, Ribeiro H, da Silva JA, Mahu I, Domingos AI, Veiga-Fernandes H. Neuro-mesenchymal units control ILC2 and obesity via a brain-adipose circuit. Nature. 2021 Sep;597(7876):410-414. doi: 10.1038/s41586-021-03830-7. Epub 2021 Aug 18. PMID 34408322
- [Background] Zeng W, Pirzgalska RM, Pereira MM, Kubasova N, Barateiro A, Seixas E, Lu YH, Kozlova A, Voss H, Martins GG, Friedman JM, Domingos AI. Sympathetic neuro-adipose connections mediate leptin-driven lipolysis. Cell. 2015 Sep 24;163(1):84-94. doi: 10.1016/j.cell.2015.08.055. PMID 26406372
- [Background] Farruggia MC, Small DM. Effects of adiposity and metabolic dysfunction on cognition: A review. Physiol Behav. 2019 Sep 1;208:112578. doi: 10.1016/j.physbeh.2019.112578. Epub 2019 Jun 11. PMID 31194997
- [Background] Gardener H, Caunca M, Dong C, Cheung YK, Rundek T, Elkind MSV, Wright CB, Sacco RL. Obesity Measures in Relation to Cognition in the Northern Manhattan Study. J Alzheimers Dis. 2020;78(4):1653-1660. doi: 10.3233/JAD-201071. PMID 33164939
- [Background] Dahl AK, Hassing LB, Fransson EI, Gatz M, Reynolds CA, Pedersen NL. Body mass index across midlife and cognitive change in late life. Int J Obes (Lond). 2013 Feb;37(2):296-302. doi: 10.1038/ijo.2012.37. Epub 2012 Mar 27. PMID 22450854
- [Background] Tang X, Zhao W, Lu M, Zhang X, Zhang P, Xin Z, Sun R, Tian W, Cardoso MA, Yang J, Simo R, Zhou JB, Stehouwer CDA. Relationship between Central Obesity and the incidence of Cognitive Impairment and Dementia from Cohort Studies Involving 5,060,687 Participants. Neurosci Biobehav Rev. 2021 Nov;130:301-313. doi: 10.1016/j.neubiorev.2021.08.028. Epub 2021 Aug 28. PMID 34464646
- [Background] Qu Y, Hu HY, Ou YN, Shen XN, Xu W, Wang ZT, Dong Q, Tan L, Yu JT. Association of body mass index with risk of cognitive impairment and dementia: A systematic review and meta-analysis of prospective studies. Neurosci Biobehav Rev. 2020 Aug;115:189-198. doi: 10.1016/j.neubiorev.2020.05.012. Epub 2020 May 30. PMID 32479774
- [Background] Endle H, Horta G, Stutz B, Muthuraman M, Tegeder I, Schreiber Y, Snodgrass IF, Gurke R, Liu ZW, Sestan-Pesa M, Radyushkin K, Streu N, Fan W, Baumgart J, Li Y, Kloss F, Groppa S, Opel N, Dannlowski U, Grabe HJ, Zipp F, Racz B, Horvath TL, Nitsch R, Vogt J. AgRP neurons control feeding behaviour at cortical synapses via peripherally derived lysophospholipids. Nat Metab. 2022 Jun;4(6):683-692. doi: 10.1038/s42255-022-00589-7. Epub 2022 Jun 27. PMID 35760867
- [Background] Suarez AN, Hsu TM, Liu CM, Noble EE, Cortella AM, Nakamoto EM, Hahn JD, de Lartigue G, Kanoski SE. Gut vagal sensory signaling regulates hippocampus function through multi-order pathways. Nat Commun. 2018 Jun 5;9(1):2181. doi: 10.1038/s41467-018-04639-1. PMID 29872139
- [Background] Minhas PS, Latif-Hernandez A, McReynolds MR, Durairaj AS, Wang Q, Rubin A, Joshi AU, He JQ, Gauba E, Liu L, Wang C, Linde M, Sugiura Y, Moon PK, Majeti R, Suematsu M, Mochly-Rosen D, Weissman IL, Longo FM, Rabinowitz JD, Andreasson KI. Restoring metabolism of myeloid cells reverses cognitive decline in ageing. Nature. 2021 Feb;590(7844):122-128. doi: 10.1038/s41586-020-03160-0. Epub 2021 Jan 20. PMID 33473210
- [Background] Coin-Araguez L, Pavon FJ, Contreras A, Gentile AM, Lhamyani S, De Diego-Otero Y, Casado Y, Oliva Olivera W, Olveira G, Tinahones FJ, Perez Costillas L, El Bekay R. Inflammatory gene expression in adipose tissue according to diagnosis of anxiety and mood disorders in obese and non-obese subjects. Sci Rep. 2018 Nov 30;8(1):17518. doi: 10.1038/s41598-018-35759-9. PMID 30504920
- [Background] Das SK, Ma L, Sharma NK. Adipose tissue gene expression and metabolic health of obese adults. Int J Obes (Lond). 2015 May;39(5):869-73. doi: 10.1038/ijo.2014.210. Epub 2014 Dec 18. PMID 25520251
- [Background] Scherer PE. Adipose tissue: from lipid storage compartment to endocrine organ. Diabetes. 2006 Jun;55(6):1537-45. doi: 10.2337/db06-0263. PMID 16731815
- [Background] Longo M, Zatterale F, Naderi J, Parrillo L, Formisano P, Raciti GA, Beguinot F, Miele C. Adipose Tissue Dysfunction as Determinant of Obesity-Associated Metabolic Complications. Int J Mol Sci. 2019 May 13;20(9):2358. doi: 10.3390/ijms20092358. PMID 31085992